CLINICAL TRIAL: NCT00987766
Title: Phase Ib Trial of Gemcitabine and Oxaliplatin (GEMOX) With Erlotinib in Patients With Advanced Biliary Tract Cancer.
Brief Title: Gemcitabine Hydrochloride, Oxaliplatin, and Erlotinib Hydrochloride in Treating Patients With Advanced Biliary Tract Cancer, Pancreatic Cancer, Duodenal Cancer, or Ampullary Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Laura W. Goff, MD, Assistant Professor of Medicine; Associate Director, Hematology/Oncology Fellowship Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 0906; P30CA068485 (NIH)
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Extrahepatic Bile Duct Cancer; Gallbladder Cancer; Liver Cancer; Pancreatic Cancer; Periampullary Adenocarcinoma; Small Intestine Cancer
Keywords: advanced adult primary liver cancer; stage III pancreatic cancer; stage IV pancreatic cancer; periampullary adenocarcinoma; small intestine adenocarcinoma; adenocarcinoma of the extrahepatic bile duct; adenocarcinoma of the gallbladder; unresectable extrahepatic bile duct cancer; unresectable gallbladder cancer
MeSH Terms: conditions — Bile Duct Neoplasms; Gallbladder Neoplasms; Liver Neoplasms; Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Gemcitabine + Oxaliplatin + Erlotinib
  Interventions: Drug: erlotinib hydrochloride; Drug: gemcitabine hydrochloride; Drug: oxaliplatin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: erlotinib hydrochloride — Taken daily by mouth for 6 days every other week.
Drug: gemcitabine hydrochloride — Given through a vein in the arm 1 time every other week.
Drug: oxaliplatin — Given through a vein in the arm 1 time every other week.
Other: laboratory biomarker analysis — Blood and tissue collection.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine hydrochloride and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving gemcitabine hydrochloride and oxaliplatin together with erlotinib hydrochloride may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of erlotinib hydrochloride when given together with gemcitabine hydrochloride and oxaliplatin in treating patients with advanced biliary tract cancer, pancreatic cancer, duodenal cancer, or ampullary cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose and the recommended phase II dose of erlotinib hydrochloride in combination with gemcitabine hydrochloride and oxaliplatin in patients with advanced biliary tract cancer, pancreatic cancer, duodenal cancer, or ampullary cancer.

Secondary

* To describe any antitumor activity associated with this treatment regimen when given during the dose-escalation and expanded-cohort portions of this study.
* To evaluate e-cadherin, vimentin, fibronectin, amphiregulin, and Kras status in the tumors and assess their relationship to response.

OUTLINE: This is a multicenter, dose-escalation study of erlotinib hydrochloride.

Patients receive gemcitabine hydrochloride IV on day 1, oxaliplatin IV over 2 hours on day 2, and oral erlotinib hydrochloride once daily on days 3-8. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.

Tumor tissue samples are collected for biomarker and other analysis.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Only advanced carcinomas defined as unresectable or metastatic that are histologically or cytologically confirmed to be biliary tract, pancreas, duodenal, or ampullary carcinomas will be included.
* Dose-escalation: Patients > 18 years of age with biopsy-confirmed advanced biliary tract adenocarcinoma, pancreas cancer, duodenal cancer, or ampullary cancer
* MTD expansion cohort: Patients > 18 years of age with biopsy-confirmed advanced biliary tract adenocarcinoma only.
* No prior chemotherapy or prior EGF receptor inhibitor therapy
* Measurable tumor by imaging examination
* Performance status (PS) 0-2 on the ECOG performance scale
* Have pretreatment bilirubin<2.5x upper limit of normal (ULN), serum creatinine<1.5x ULN, AST and ALT <2.5xULN or in the presence of liver metastasis <5xULN, neutrophils>1500, platelets>100K, hemoglobin >9 g/dL
* Patients - both males and females - with reproductive potential (ie, menopausal for less than 1 year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration.
* Have the ability to understand the requirements of the study and provide informed consent

Exclusion Criteria:

* CNS metastases
* Uncontrolled infection
* Pregnant or nursing women may not participate.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.
* Psychiatric illness that would prevent understanding the nature of the investigational therapy and complying with protocol requirements
* Patients with > grade 2 neuropathy
* Patients with > grade 2 uncontrolled nausea and vomiting despite antiemetics
* Any concurrent medical condition that, in the judgment of the investigator, would make the patient an inappropriate candidate for study enrollment
* Prior chemotherapy or EGFR inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-11; Primary Completion 2013-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose and recommended phase II dose of erlotinib hydrochloride in combination with gemcitabine hydrochloride and oxaliplatin | 28 days

SECONDARY OUTCOMES:
Antitumor activity | 30 days after completing treatment.
E-cadherin, vimentin, fibronectin, amphiregulin, and Kras status in the tumors and their relationship to response | 30 days after completing treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Goff, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/